CLINICAL TRIAL: NCT03560128
Title: Comparison of Endocuff Vision to Medivators AmplifEYE for Detection of Precancerous Colorectal Polyps.
Brief Title: Endocuff Vision Colonoscopy vs. AmplifEYE Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1802193017
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Adenoma; Colorectal Polyp; Colorectal Cancer
Keywords: Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Endocuff Vision Arm (Experimental): Colonoscopy with Endocuff Vision device attached to the distal end of the scope.
  Interventions: Device: Endocuff Vision device
- AmplifEYE Arm (Experimental): Colonoscopy with AmplifEYE device attached to the distal end of the scope.
  Interventions: Device: AmplifEYE device

INTERVENTIONS:
Device: Endocuff Vision device — Subjects randomized to undergo a colonoscopy procedure with the Endocuff Vision device will have this device placed on the colonoscope used during their procedure.
  Arms: Endocuff Vision Arm
Device: AmplifEYE device — Subjects randomized to undergo a colonoscopy procedure with the AmplifEYE device will have this device placed on the colonoscope used during their procedure.
  Arms: AmplifEYE Arm

SUMMARY:
The study aims to compare the results between colonoscopies with two different attachments on the distal end of the colonoscope.

DETAILED DESCRIPTION:
This will be a prospective, randomized controlled study. Subjects referred for a screening, surveillance, or diagnostic colonoscopy will be prospectively enrolled. This study aims to compare the number of adenomas detected per colonoscopy (APC) between an Endocuff colonoscopy and an AmplifEYE colonoscopy.

It is estimated that the Endocuff Vision will result in an APC of 2.3. The investigators consider that a clinically acceptable ADR for the Medivators device would be within 20% of this value or 1.5.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Undergoing colonoscopy for screening, surveillance, or diagnostic purposes
* Able to provide written informed consent

Exclusion Criteria:

* Active Inflammatory Bowel Disease
* Prior resection of the colon
* Referred for resection of a polyp identified by another physician
* Referred for a previous incomplete colonoscopy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data can be shared in the future upon request.

REFERENCES:
- [Background] Rex DK, Repici A, Gross SA, Hassan C, Ponugoti PL, Garcia JR, Broadley HM, Thygesen JC, Sullivan AW, Tippins WW, Main SA, Eckert GJ, Vemulapalli KC. High-definition colonoscopy versus Endocuff versus EndoRings versus full-spectrum endoscopy for adenoma detection at colonoscopy: a multicenter randomized trial. Gastrointest Endosc. 2018 Aug;88(2):335-344.e2. doi: 10.1016/j.gie.2018.02.043. Epub 2018 Mar 9. PMID 29530353
- [Derived] Rex DK, Sagi SV, Kessler WR, Rogers NA, Fischer M, Bohm ME, Dewitt JM, Lahr RE, Searight MP, Sullivan AW, McWhinney CD, Garcia JR, Broadley HM, Vemulapalli KC. A comparison of 2 distal attachment mucosal exposure devices: a noninferiority randomized controlled trial. Gastrointest Endosc. 2019 Nov;90(5):835-840.e1. doi: 10.1016/j.gie.2019.06.046. Epub 2019 Jul 15. PMID 31319060

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Started | 306 | 306
Completed | 294 | 298
Not Completed | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm | Total
Number analyzed (Participants) | 294 | 298 | 592
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10) | 63.2 (9.7) | 62.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 170 | 325
  Male | 139 | 128 | 267
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 264 | 268 | 532
  Other | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 294 | 298 | 592
Indication for Procedure [Count of Participants; unit: Participants]
  Screening | 100 | 113 | 213
  Diagnostic | 18 | 24 | 42
  Surveillance | 171 | 160 | 331

OUTCOME MEASURES:

1. Primary Outcome: Number of Adenomas Detected Per Colonoscopy (APC).
Description: Comparison of the number of adenomas detected per colonoscopy between the Endocuff Vision Colonoscopy and the AmplifEYE colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Mean (Standard Deviation); unit: adenomas
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
adenomas | 1.63 (2.8) | 1.51 (2.3)

2. Secondary Outcome: Detection Rates (Adenoma Detection Rate (ADR) and Polyp Detection Rate (PDR))
Description: Comparison of the number of participants with at least one adenoma detected (ADR) between AmplifEYE colonoscopy and the Endocuff Vision colonoscopy.
  Comparison of the number of participants with at least one polyp detected (PDR) between AmplifEYE colonoscopy and the Endocuff Vision colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
Participants
  at least 1 detected adenoma | 164 | 159
  at least 1 detected polyp | 229 | 231

3. Secondary Outcome: Complications Encountered During Procedure
Description: Comparison of amount of mucosal trauma (such as scratches), perforation (making a hole in the colon wall), or gastrointestinal bleeding between patients that have AmplifEYE colonoscopy compared to patients that have Endocuff Vision colonoscopy.
Time Frame: During Colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
Participants
  Mucosal Trauma | 30 | 24
  GI Bleeding | 0 | 0
  Perforation | 0 | 0

4. Secondary Outcome: Passage of Device Through Sigmoid Colon
Description: Comparison of the number of times the device had to be removed to pass the sigmoid colon between colonoscopies with the AmplifEYE device and colonoscopies with the Endocuff Vision device.
Time Frame: during insertion portion of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
Participants | 17 | 15

5. Secondary Outcome: Polyps Per Colonoscopy (PPC)
Description: Comparison of the number of polyps detected per colonoscopy between the Endocuff Vision Colonoscopy and the AmplifEYE colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Mean (Standard Deviation); unit: Polyps
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
Polyps | 2.71 (3.4) | 2.55 (2.9)

6. Secondary Outcome: Time Comparison for Each Method
Description: Comparison of the insertion time, overall withdrawal time, inspection time, and total procedure time between the AmplifEYE colonoscopy and the Endocuff Vision colonoscopy.
  Insertion time: time it takes from the colonoscope first being inserted to when the cecum is reached Withdrawal time: time calculated from when withdrawing is started in the cecum until the colonoscope is removed. This includes time spent washing, suctioning, inspecting the colon, and removing polyps.
  Inspection time: time spent actually examining the colon and does not include time spent for washing the colon, suctioning, and removing polyps.
  Total procedure time: time from the initial insertion of the colonoscope through the complete withdrawal of the colonoscope.
Time Frame: During colonoscopy procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
Minutes
  Insertion Time | 5.6 (3.7) | 5.7 (4.1)
  Overall Withdrawal Time | 14.6 (6.2) | 14.9 (6.3)
  Inspection Time | 6.8 (2.3) | 6.9 (1.6)
  Total Procedure Time | 21.1 (7.8) | 21.5 (7.6)

7. Secondary Outcome: Cecal Intubation Rate
Description: Comparison of the number of procedures where the colonoscope was able to reach the cecum between AmplifEYE colonoscopy and Endocuff Vision colonoscopy.
Time Frame: During Colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
Participants | 294 | 297

8. Secondary Outcome: Detection of Serrated Lesions
Description: Comparison of the number of participants with at least one Sessile Serrated Polyp detected (SSPDR) between AmplifEYE colonoscopy and the Endocuff Vision colonoscopy.
  Comparison of the number of participants with at least one flat polyp detected between AmplifEYE colonoscopy and the Endocuff Vision colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
Number analyzed (Participants) | 294 | 298
Participants
  at least one sessile serrated polyp detected | 40 | 46
  at least one flat polyp detected | 122 | 130

ADVERSE EVENTS:
Time Frame: During the colonoscopy procedure until the time the patient left the endoscopy suite.
Arm/Group | AmplifEYE Arm | Endocuff Vision Arm
All-Cause Mortality (participants affected / at risk) | 0/294 | 0/298
Serious Adverse Events (participants affected / at risk) | 0/294 | 0/298
Other Adverse Events (participants affected / at risk) | 0/294 | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03560128/Prot_SAP_000.pdf